CLINICAL TRIAL: NCT06512376
Title: Hereditary Cerebral Small Vessel Diseases Registry-Trial Ready Cohort (HCSVD-TRC)
Brief Title: Hereditary Cerebral Small Vessel Diseases Registry-Trial Ready Cohort
Acronym: HCSVD-TRC
Status: Active, not recruiting | Type: Observational
Sponsor: Beijing Tiantan Hospital (Other)
Responsible Party: Principal Investigator, yilong Wang, Vice President of Beijing Tiantan Hospital, Beijing Tiantan Hospital
Other Study IDs: KY-2022-074-02
Record Dates: First submitted 2024-07-16; First posted 2024-07-22 (Actual); Last update posted 2024-07-22 (Actual); Status verified 2024-01

CONDITIONS: Cerebral Small Vessel Diseases; Hereditary
Keywords: hCSVD; multi-center; prospective; continuous; registry
MeSH Terms: conditions — Cerebral Small Vessel Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 5 Years
Biospecimen Retention: Samples With DNA — Blood and urine samples will be collected at baseline, 6 months, 1 year, 2 years, 3 years, 4 years, and 5 years to test genetic and metabolomic markers.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
We took hereditary cerebral small vessel disease (hCSVD) patients as our main subjects, aiming to establish a platform for a comprehensive evaluation and long-term follow-up. Deeply explore the pathophysiological mechanism of hCSVD, which may render the theoretical basis for the treatment and management of hCSVD.

DETAILED DESCRIPTION:
Cerebral Small Vessel Disease is a series of clinical, imaging, and pathological syndromes caused by a variety of risk factors affecting cerebral arterioles, arterioles, capillaries, and venules, accounting for 20% of stroke and 45% of dementia.

Although the incidence rate of hereditary small cerebral vascular disease is low, because of its early onset, high disability rate, and lack of effective treatment, it also brings a heavy burden to the patients and their families. Therefore, it is important to study the pathogenic gene, pathogenesis, clinical characteristics, and imaging manifestations of hereditary cerebrovascular disease to provide a theoretical basis for the treatment and prevention of hereditary cerebrovascular disease in the future.

This multi-center, prospective, continuous, registry study, runs from 2022 to 2027. The study is expected to recruit 100 subjects, according to the sample size design of the registry study.

We recruited patients with the hereditary cerebral small-vessel disease (hCSVD) intending to establish a platform for a comprehensive assessment and long-term follow-up by collecting genetics, imaging, and clinical symptoms of the primary disease and its relatives. With long-term follow-up of the development and prognosis of imaging and clinical symptoms combined with genetics, we will work on the correlation between genes and phenotype and deeply explore the pathophysiological mechanism of hCSVD, which may render the theoretical basis for the treatment and management of hCSVD.

ELIGIBILITY:
Inclusion Criteria:

1. All ages, male or female
2. Carriers of the pathogenic genes mutation (mutation with unknown clinical significance/ suspected pathogenic mutation/ pathogenic mutation) of hCSVD confirmed by the gene tests, including but not limited to NOTCH3, HTPA1, CTSA, GLA, TREX1, COL4A1/2, or highly-suspected hCSVD2
3. CSVD related abnormalities on brain MRI, any 1 or more of:

   1. White matter hyperintensities, Fazekas score3 ≥1
   2. ≥1 newly-occurred lacunar infarcts
   3. ≥1 old lacunar infarcts
   4. ≥3 cerebral microbleeds
4. Informed consent signed

Exclusion Criteria:

1. Diagnosis of mental disorders according to DSM-V and unable to be compliant to the research
2. Patients with life expectancy less than one year due to any advanced disease, e.g., malignant tumor
3. Patients unable to return for follow-up visits due to some reasons

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: hCSVD with identified gene mutations, and highly-suspected hCSVD without any identified gene mutation
Sampling Method: Non-Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2022-07-19 (Actual); Primary Completion 2027-07-19 (Estimated); Study Completion 2027-07-19 (Estimated)

PRIMARY OUTCOMES:
The epidemiological features | at baseline
  Any epidemiological informations
The clinical features | 5 years
  Clinical symptoms and physical examination
The radiography features | at baseline
  Neuroimaging markers collected by MRI
A novel pathogenic gene for hereditary cerebrovascular disease in the Chinese population | at baseline
  Genetic testing with the blood sample

SECONDARY OUTCOMES:
Etiology and pathogenesis | at baseline
  This study will collect etiology and pathogenesis information among participants.
Long-term changes of radiography features | 5 years
  Neuroimaging markers collected by MRI

CONTACTS AND LOCATIONS:
Overall Officials: Yilong Wang, MD+PhD, Principal Investigator — Capital Medical University
Locations (1):
- Beijing Tiantan Hospital, Beijing, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Pantoni L. Cerebral small vessel disease: from pathogenesis and clinical characteristics to therapeutic challenges. Lancet Neurol. 2010 Jul;9(7):689-701. doi: 10.1016/S1474-4422(10)70104-6. PMID 20610345
- [Result] Gorelick PB, Scuteri A, Black SE, Decarli C, Greenberg SM, Iadecola C, Launer LJ, Laurent S, Lopez OL, Nyenhuis D, Petersen RC, Schneider JA, Tzourio C, Arnett DK, Bennett DA, Chui HC, Higashida RT, Lindquist R, Nilsson PM, Roman GC, Sellke FW, Seshadri S; American Heart Association Stroke Council, Council on Epidemiology and Prevention, Council on Cardiovascular Nursing, Council on Cardiovascular Radiology and Intervention, and Council on Cardiovascular Surgery and Anesthesia. Vascular contributions to cognitive impairment and dementia: a statement for healthcare professionals from the american heart association/american stroke association. Stroke. 2011 Sep;42(9):2672-713. doi: 10.1161/STR.0b013e3182299496. Epub 2011 Jul 21. PMID 21778438
- [Result] Nam KW, Kwon HM, Lim JS, Han MK, Nam H, Lee YS. The presence and severity of cerebral small vessel disease increases the frequency of stroke in a cohort of patients with large artery occlusive disease. PLoS One. 2017 Oct 9;12(10):e0184944. doi: 10.1371/journal.pone.0184944. eCollection 2017. PMID 28991905
- [Result] Federico A, Di Donato I, Bianchi S, Di Palma C, Taglia I, Dotti MT. Hereditary cerebral small vessel diseases: a review. J Neurol Sci. 2012 Nov 15;322(1-2):25-30. doi: 10.1016/j.jns.2012.07.041. Epub 2012 Aug 4. PMID 22868088
- [Result] Tan R, Traylor M, Rutten-Jacobs L, Markus H. New insights into mechanisms of small vessel disease stroke from genetics. Clin Sci (Lond). 2017 Apr 1;131(7):515-531. doi: 10.1042/CS20160825. PMID 28302914
- [Result] Adib-Samii P, Brice G, Martin RJ, Markus HS. Clinical spectrum of CADASIL and the effect of cardiovascular risk factors on phenotype: study in 200 consecutively recruited individuals. Stroke. 2010 Apr;41(4):630-4. doi: 10.1161/STROKEAHA.109.568402. Epub 2010 Feb 18. PMID 20167921
- [Result] Singhal S, Bevan S, Barrick T, Rich P, Markus HS. The influence of genetic and cardiovascular risk factors on the CADASIL phenotype. Brain. 2004 Sep;127(Pt 9):2031-8. doi: 10.1093/brain/awh223. Epub 2004 Jun 30. PMID 15229130
- [Result] de Boer I, Pelzer N, Terwindt G. Retinal Vasculopathy with Cerebral Leukoencephalopathy and Systemic Manifestations. 2019 Sep 19. In: Adam MP, Bick S, Mirzaa GM, Pagon RA, Wallace SE, Amemiya A, editors. GeneReviews(R) [Internet]. Seattle (WA): University of Washington, Seattle; 1993-2026. Available from http://www.ncbi.nlm.nih.gov/books/NBK546576/ PMID 31536185
- [Result] Mancuso M, Arnold M, Bersano A, Burlina A, Chabriat H, Debette S, Enzinger C, Federico A, Filla A, Finsterer J, Hunt D, Lesnik Oberstein S, Tournier-Lasserve E, Markus HS. Monogenic cerebral small-vessel diseases: diagnosis and therapy. Consensus recommendations of the European Academy of Neurology. Eur J Neurol. 2020 Jun;27(6):909-927. doi: 10.1111/ene.14183. Epub 2020 Mar 20. PMID 32196841
- [Result] Peters N, Freilinger T, Opherk C, Pfefferkorn T, Dichgans M. Effects of short term atorvastatin treatment on cerebral hemodynamics in CADASIL. J Neurol Sci. 2007 Sep 15;260(1-2):100-5. doi: 10.1016/j.jns.2007.04.015. Epub 2007 May 24. PMID 17531269
- [Result] Germain DP, Charrow J, Desnick RJ, Guffon N, Kempf J, Lachmann RH, Lemay R, Linthorst GE, Packman S, Scott CR, Waldek S, Warnock DG, Weinreb NJ, Wilcox WR. Ten-year outcome of enzyme replacement therapy with agalsidase beta in patients with Fabry disease. J Med Genet. 2015 May;52(5):353-8. doi: 10.1136/jmedgenet-2014-102797. Epub 2015 Mar 20. PMID 25795794
- [Result] Schiffmann R, Kopp JB, Austin HA 3rd, Sabnis S, Moore DF, Weibel T, Balow JE, Brady RO. Enzyme replacement therapy in Fabry disease: a randomized controlled trial. JAMA. 2001 Jun 6;285(21):2743-9. doi: 10.1001/jama.285.21.2743. PMID 11386930
- [Result] Germain DP, Hughes DA, Nicholls K, Bichet DG, Giugliani R, Wilcox WR, Feliciani C, Shankar SP, Ezgu F, Amartino H, Bratkovic D, Feldt-Rasmussen U, Nedd K, Sharaf El Din U, Lourenco CM, Banikazemi M, Charrow J, Dasouki M, Finegold D, Giraldo P, Goker-Alpan O, Longo N, Scott CR, Torra R, Tuffaha A, Jovanovic A, Waldek S, Packman S, Ludington E, Viereck C, Kirk J, Yu J, Benjamin ER, Johnson F, Lockhart DJ, Skuban N, Castelli J, Barth J, Barlow C, Schiffmann R. Treatment of Fabry's Disease with the Pharmacologic Chaperone Migalastat. N Engl J Med. 2016 Aug 11;375(6):545-55. doi: 10.1056/NEJMoa1510198. PMID 27509102
- [Result] Rutten JW, Dauwerse HG, Peters DJ, Goldfarb A, Venselaar H, Haffner C, van Ommen GJ, Aartsma-Rus AM, Lesnik Oberstein SA. Therapeutic NOTCH3 cysteine correction in CADASIL using exon skipping: in vitro proof of concept. Brain. 2016 Apr;139(Pt 4):1123-35. doi: 10.1093/brain/aww011. Epub 2016 Feb 19. PMID 26912635
- [Result] Liu XY, Gonzalez-Toledo ME, Fagan A, Duan WM, Liu Y, Zhang S, Li B, Piao CS, Nelson L, Zhao LR. Stem cell factor and granulocyte colony-stimulating factor exhibit therapeutic effects in a mouse model of CADASIL. Neurobiol Dis. 2015 Jan;73:189-203. doi: 10.1016/j.nbd.2014.09.006. Epub 2014 Sep 22. PMID 25251607